CLINICAL TRIAL: NCT00718965
Title: A Double-blind, Randomized, 12-month, Placebo-controlled, Parallel Group, Fixed-dose Study to Evaluate the Efficacy and Safety of AVE5530 25mg/Day and AVE5530 50 mg/Day in Patients With Primary Hypercholesterolemia
Brief Title: Evaluation of Efficacy and Safety of AVE5530 in Patients With Primary Hypercholesterolemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: AVE5530 in hypercholesterolemia was stopped due to insufficient efficacy
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC6909
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Hypercholesterolemia
Keywords: Primary hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 25 mg/day AVE5530 (Experimental)
  Interventions: Drug: AVE5530
- 50 mg/day AVE5530 (Experimental)
  Interventions: Drug: AVE5530
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVE5530 — one tablet in the evening with dinner
  Arms: 25 mg/day AVE5530; 50 mg/day AVE5530
Drug: Placebo — one tablet in the evening with dinner
  Arms: Placebo

SUMMARY:
The present study is aiming at assessing the efficacy and safety of AVE5530 (25mg and 50mg) in a double-blind comparison with placebo in the management of patients with primary hypercholesterolemia. The main objective is to evaluate the effects of AVE5530 on LDL-C level reduction as adjunct to a controlled diet. The effects of AVE5530 on other lipid parameters will be assessed as secondary objectives.

DETAILED DESCRIPTION:
The study will include a 2-week pre-randomization placebo lead-in phase and a double-blind treatment period of at least 12 months and can be variably extended up to approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults with high cholesterol levels either not receiving or willing and able to discontinue ongoing lipid-lowering therapy

Exclusion Criteria:

* LDL-C levels > 250 mg/dL (6.48 mmol/L)
* Triglycerides levels > 350mg/dL (3.95 mmol/L)
* Conditions / situations such as:

  * presence of any clinically significant uncontrolled endocrine disease known to influence lipids levels
  * Active liver disease
  * High estimated risk of Coronary Heart Disease
  * Recent history of congestive heart failure , of unstable angina pectoris, myocardial infarction, coronary bypass surgery or angioplasty, or Unstable or severe peripheral artery disease
  * Positive test for Hepatitis B surface antigen and/or Hepatitis C antibody or Known to be Human Immunodeficient Virus (HIV) positive
* Pregnant or breast-feeding women,
* Women of childbearing potential not protected by effective contraceptive method of birth control (including oral contraceptives) and/or who are unwilling or unable to be tested for pregnancy prior to exposure to the Investigational Product.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 826 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
percent change from baseline in calculated LDL-C | at week 12

SECONDARY OUTCOMES:
percent change from baseline in calculated LDL-C | at 6 months and 12 months
percent change from baseline in total cholesterol and Apo-B | at 12 weeks, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John CROUSE, MD, Principal Investigator — Wake Forest University Health Sciences, North Carolina, US
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, San Juan, Puerto Rico